CLINICAL TRIAL: NCT06777641
Title: Development and Assessment of a Point-of-Care Ultrasound (PoCUS) Low-Contact Curriculum Using Near-Peer Training and Remote Supervision
Brief Title: Point-of-Care Ultrasound (PoCUS) Low-Contact Curriculum Using Near-Peer Training and Remote Supervision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Clinical Trial Center (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, NTUH-CTC, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 202410061RINE
Record Dates: First submitted 2025-01-10; First posted 2025-01-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-01

CONDITIONS: Educational Problems
Keywords: ultrasound; peer teaching; remote supervision

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): This group will experience lectures combined with peer instructor for hands-on training (lecture + NPT hands-on with remote supervision). The PoCUS teacher will not be physically present but will supervise remotely via video conferencing to monitor and communicate in real-time.
  Interventions: Other: remote supervision
- Control (No Intervention): This group will follow the conventional teaching model, combining lectures with on-site PoCUS teacher supervised hands-on training (lecture + on-site teacher supervised hands-on).

INTERVENTIONS:
Other: remote supervision — teacher use remote supervision to assist peer training
  Arms: Experimental

SUMMARY:
Ultrasonography is a non-invasive, minimal-radiation tool for clinical diagnosis. Relevant clinical protocols have been developed. Recently, as the technology of ultrasonography progresses, small and portable ultrasound machines become available. The use of ultrasonography has gradually moved from the examination laboratories to the bedside. With this revolution, ultrasonography produces a tremendous paradigm shift in the diagnostic process at the bedside by clinicians. Point-of-care ultrasound (PoCUS) focuses on an acute problem that a patient has, trying to simplify the items of examination, shorten the time required for examination, but maximize the efficiency and accessibility. Unlike traditional ultrasound which has high learning threshold, PoCUS has become a feasible curriculum for undergraduate medical students and also post-graduate residents. However, the needs assessment, curriculum design, assessment tools of PoCUS education for medical students are scarcely reported. And the effectiveness of using new teaching skills, such as E-learning, standardized patient simulation, and high-fidelity simulators, in teaching PoCUS remains unanswered. There is also no established assessment tool for learning PoCUS in undergraduate medical education.

The COVID-19 pandemic also challenges medical education, including the training of PoCUS. As a skill-based curriculum, a pure E-learning is not feasible. Therefore, an important issue is to find a way to lower the physical contact during the PoCUS training. To date, scarce study has focused on the contact time and contact density of a skill-based curriculum. The main purpose of this study is establishing a low-contact PoCUS curriculum, with incorporation of small group teaching, near-peer training (NPT) design, and remote supervision (RS). It is also mandatory to make sure the effectiveness of this new curriculum, through a competency-based assessment such as entrustable professional activity (EPA). In the second year of the project, students will be randomized into two groups, including NPT+ RS group and traditional groups, to compare the amount and intensity of contact during curriculum and the effectiveness of training through objective structured clinical examination (OSCE) between two groups.

DETAILED DESCRIPTION:
Background Ultrasonography is a non-invasive, minimal-radiation tool for clinical diagnosis. Relevant clinical protocols have been developed. Recently, as the technology of ultrasonography progresses, small and portable ultrasound machines become available. The use of ultrasonography has gradually moved from the examination laboratories to the bedside. With this revolution, ultrasonography produces a tremendous paradigm shift in the diagnostic process at the bedside by clinicians. Point-of-care ultrasound (PoCUS) focuses on an acute problem that a patient has, trying to simplify the items of examination, shorten the time required for examination, but maximize the efficiency and accessibility. Unlike traditional ultrasound which has high learning threshold, PoCUS has become a feasible curriculum for undergraduate medical students and also post-graduate residents. However, the needs assessment, curriculum design, assessment tools of PoCUS education for medical students are scarcely reported. And the effectiveness of using new teaching skills, such as E-learning, standardized patient simulation, and high-fidelity simulators, in teaching PoCUS remains unanswered. There is also no established assessment tool for learning PoCUS in undergraduate medical education.

The COVID-19 pandemic also challenges medical education, including the training of PoCUS. As a skill-based curriculum, a pure E-learning is not feasible. Therefore, an important issue is to find a way to lower the physical contact during the PoCUS training. Traditional PoCUS courses involve direct teaching by instructors, with students attending lectures and practicing hands-on ultrasound or simulator skills during the second half of the course. This teaching model, combining didactic lectures and hands-on practice, is internationally recognized as effective. Some studies even suggest that hands-on sessions should comprise at least 50% of the total course time. While this method yields excellent learning outcomes, it involves close and prolonged contact between instructors and students, posing a high risk of infection transmission, making it unsuitable during the COVID-19 pandemic.

To date, scarce study has focused on the contact time and contact density of a skill-based curriculum. The main purpose of this study is establishing a low-contact PoCUS curriculum, with incorporation of small group teaching, near-peer training (NPT) design, and remote supervision (RS).

Material and Methods Similar to the Resident as Teacher (RaT) model promoted in other medical education fields, student teachers leading peer training in Near-Peer Teaching (NPT) must undergo training before their formal teaching sessions. During the first phase of the plan, medical students and residents volunteering as peer instructors participated in trial teaching sessions under observation, with faculty sitting in the audience to evaluate. After each session, the faculty provided immediate feedback and assessed whether these seed teachers were qualified to take on the role of NPT instructors in the second-phase plan.

To enable remote supervision by faculty, it was essential to ensure an unobstructed view of the on-site activities during skill sessions. Camera angles were determined to cover critical perspectives. Ideally, 2-3 cameras are necessary to provide a comprehensive view for remote supervision. The cameras must capture the following: (1)Ultrasound Screen: The ultrasound images displayed on the machine; (2)Operator's Hands and Probe Placement: The hand gestures of the student holding the ultrasound probe and its placement on the patient's body. After pilot testing in the first phase, video recordings of the sessions were reviewed during expert meetings to refine the setup. This process informed the design of the second-year comparative study and the calculation of contact density from the videos.

The study assumes that remote supervision reduces direct contact between teachers and students. However, the contact between seed student teachers and learners will be assessed through recorded footage and expert discussion. Since similar studies do not exist for reference, the primary endpoint of this research is learning outcomes, with contact density as a secondary endpoint.

In the second phase, medical students in their fifth or sixth year will be recruited through poster advertisements for voluntary participation. After inform consent, the participating medical students will be randomly assigned to two groups:

1. Traditional Group (Control Group): This group will follow the conventional teaching model, combining lectures with on-site PoCUS teacher supervised hands-on training (lecture + on-site teacher supervised hands-on).
2. Experimental Group: This group will experience lectures combined with peer instructor for hands-on training (lecture + NPT hands-on with remote supervision). The PoCUS teacher will not be physically present but will supervise remotely via video conferencing to monitor and communicate in real-time.

Inclusion and Exclusion Criteria:

Inclusion Criteria:

1. Fifth- or sixth-year medical students at National Taiwan University College of Medicine, aged 20 or older.

Exclusion Criteria:

1. Unwillingness to participate in the study.
2. Prior exposure to the bedside ultrasound course at National Taiwan University College of Medicine.

To allow comparison, 80 fifth or sixth year medical students will be recruited. Participation is voluntary, and students who opt out will still have the opportunity to attend related PoCUS courses offered by the medical school. However, only students who have not previously taken a bedside ultrasound course will be eligible for this study. Students unwilling to participate in the study will also be excluded.

The inclusion of students will be voluntary, conducted under fair and open conditions without psychological pressure. Participation or non-participation in the study will not affect their grades or job performance evaluations. Students who decline to participate will receive the same course as those who agree to participate.

Endpoints Learners' feedback on the new curriculum, using the Technology Acceptance Model (TAM) will be collected after the PoCUS course and before the OSCE testing. The effectiveness of the curriculum will be evaluated approximately one month after completing the PoCUS course for both the experimental and control groups, using OSCE assessments incorporating EPA constructs. The OSCE will be evaluated independently by two reviewers, with the final score calculated as the average of their individual assessments. Students' performance will be analyzed based on their total OSCE scores as well as their scores for each construct of the EPA.

After the OSCE, a survey on the feedback on OSCE test will also be conducted.

Conclusion:

This project aims to develop a low-contact point-of-care ultrasound (PoCUS) course tailored for healthcare settings during a pandemic. It will compare the effectiveness of the new curriculum with traditional methods in reducing contact time and density during the course.

The teaching course will utilize near-peer training (NPT) combined with remote supervision through real-time video conferencing and multi-camera setups. The project seeks to verify that the new low-contact teaching model is non-inferior to the traditional method in terms of learning outcomes while significantly reducing the risk of contact-based infection.

The anticipated results will serve as valuable references for conducting effective skill teaching during pandemic conditions.

ELIGIBILITY:
Inclusion Criteria:

■Fifth- or sixth-year medical students at National Taiwan University College of Medicine, aged 20 or older.

Exclusion Criteria:

* Unwillingness to participate in the study.
* Prior exposure to the bedside ultrasound course at National Taiwan University College of Medicine.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance score on OSCE | 1 month
  The effectiveness of the curriculum will be evaluated approximately one month after completing the PoCUS course for both the experimental and control groups, using OSCE assessments incorporating EPA constructs. The OSCE will be evaluated independently by two reviewers, with the final score calculated as the average of their individual assessments. Students' performance will be analyzed based on their total OSCE scores as well as their scores for each construct of the EPA.

SECONDARY OUTCOMES:
TAM survey | 1 month
  Learners' feedback on the new curriculum, using the Technology Acceptance Model (TAM) will be collected after the PoCUS course and before the OSCE testing.
Survey of OSCE test | 1 month
  After the OSCE, a survey on the feedback on OSCE test will also be conducted.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) regarding the survey of TAM model and feedbak on OSCE test will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of the study
Access Criteria: Upon request to the principal investigator with relevant IRB consent

REFERENCES:
- [Background] ten Cate O. Entrustability of professional activities and competency-based training. Med Educ. 2005 Dec;39(12):1176-7. doi: 10.1111/j.1365-2929.2005.02341.x. No abstract available. PMID 16313574
- [Background] Frenk J, Chen L, Bhutta ZA, Cohen J, Crisp N, Evans T, Fineberg H, Garcia P, Ke Y, Kelley P, Kistnasamy B, Meleis A, Naylor D, Pablos-Mendez A, Reddy S, Scrimshaw S, Sepulveda J, Serwadda D, Zurayk H. Health professionals for a new century: transforming education to strengthen health systems in an interdependent world. Lancet. 2010 Dec 4;376(9756):1923-58. doi: 10.1016/S0140-6736(10)61854-5. Epub 2010 Nov 26. No abstract available. PMID 21112623
- [Background] Lichtenstein D, Malbrain ML. Critical care ultrasound in cardiac arrest. Technological requirements for performing the SESAME-protocol--a holistic approach. Anaesthesiol Intensive Ther. 2015;47(5):471-81. doi: 10.5603/AIT.a2015.0072. Epub 2015 Nov 18. PMID 26578398
- [Background] Lichtenstein DA, Meziere GA. Relevance of lung ultrasound in the diagnosis of acute respiratory failure: the BLUE protocol. Chest. 2008 Jul;134(1):117-25. doi: 10.1378/chest.07-2800. Epub 2008 Apr 10. PMID 18403664
- [Background] Shokoohi H, Boniface KS, Zaragoza M, Pourmand A, Earls JP. Point-of-care ultrasound leads to diagnostic shifts in patients with undifferentiated hypotension. Am J Emerg Med. 2017 Dec;35(12):1984.e3-1984.e7. doi: 10.1016/j.ajem.2017.08.054. Epub 2017 Aug 26. PMID 28851498
- [Background] Kirkpatrick AW, Sirois M, Laupland KB, Liu D, Rowan K, Ball CG, Hameed SM, Brown R, Simons R, Dulchavsky SA, Hamiilton DR, Nicolaou S. Hand-held thoracic sonography for detecting post-traumatic pneumothoraces: the Extended Focused Assessment with Sonography for Trauma (EFAST). J Trauma. 2004 Aug;57(2):288-95. doi: 10.1097/01.ta.0000133565.88871.e4. PMID 15345974
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104